CLINICAL TRIAL: NCT00012363
Title: Gemcitabine Plus Irinotecan in Patients With Esophageal Cancer, Phase II
Brief Title: S0101 Gemcitabine and Irinotecan in Treating Patients With Metastatic or Recurrent Cancer of the Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068515; S0101 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine + Irinotecan (Experimental): Gemcitabine 1000mg/m2 IV over 30 min on Days 1,8 q21days; Irinotecan 100mg/m2 IV over 90 min on Days 1,8 q21days
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: gemcitabine hydrochloride — 1,000mg/m2, IV over 30 min, days 1 & 8, q 21 days
  Other Names: Gemzar (NSC-613327)
Drug: irinotecan hydrochloride — 100 mg/m2, IV over 90 min, days 1 & 8, q 21days
  Other Names: CPT-11 (NSC-616348)

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have metastatic or recurrent cancer of the esophagus.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 6-month survival rate of patients with metastatic or recurrent carcinoma of the esophagus or gastroesophageal junction treated with gemcitabine and irinotecan.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.

OUTLINE: Patients receive gemcitabine IV over 30 minutes and irinotecan IV over 90 minutes on days 1 and 8. Treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 30-55 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic or recurrent carcinoma of the esophagus or gastroesophageal junction

  * Squamous cell carcinoma OR
  * Adenocarcinoma
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 100

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine no greater than 1.5 times upper limit of normal

Cardiovascular:

* No uncontrolled hypertension
* No unstable angina
* No symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* No serious uncontrolled cardiac arrhythmia

Gastrointestinal:

* No active inflammatory bowel disease
* No significant bowel obstruction
* No chronic diarrhea

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active infection requiring systemic therapy
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 28 days since prior biologic therapy
* No prior biologic therapy for metastatic or recurrent disease
* No concurrent sargramostim (GM-CSF)
* No concurrent immunotherapy for tumor

Chemotherapy:

* At least 28 days since prior chemotherapy
* No prior chemotherapy for metastatic or recurrent disease
* No prior gemcitabine or irinotecan
* Prior adjuvant or neoadjuvant chemotherapy at time of initial diagnosis of localized disease allowed
* No other concurrent chemotherapy for tumor

Endocrine therapy:

* See Disease Characteristics
* At least 28 days since prior endocrine therapy
* No prior endocrine therapy for metastatic or recurrent disease
* No concurrent hormonal therapy for tumor

Radiotherapy:

* At least 28 days since prior radiotherapy
* No prior radiotherapy for metastatic or recurrent disease
* Prior adjuvant or neoadjuvant radiotherapy at time of initial diagnosis of localized disease allowed
* No concurrent radiotherapy for tumor

Surgery:

* Prior thoraco-abdominal surgery allowed
* At least 3 weeks since prior surgery and recovered

Other:

* No other concurrent anti-cancer therapy for tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2001-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
6-month survival rate | 6 months after registration
  To assess the six-month survival rate in patients with esophageal cancer treated with a gemcitabine-irinotecan combination chemotherapy regimen.

SECONDARY OUTCOMES:
Toxicities | Week 1 and Week 2 of each cycle
  To assess the qualitative and quantitative toxicities associated with this regimen in a Phase II study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K. Williamson, MD, Study Chair — University of Kansas
Locations (96):
- United States (96):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP-Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - OHSU Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Result] Williamson SK, McCoy SA, Gandara DR, Dakhil SR, Yost KJ, Paradelo JC, Atkins JN, Blanke CD, Abbruzzese JL; Southwest Oncology Group (SWOG). Phase II trial of gemcitabine plus irinotecan in patients with esophageal cancer: a Southwest Oncology Group (SWOG) trial. Am J Clin Oncol. 2006 Apr;29(2):116-22. doi: 10.1097/01.coc.0000199883.10685.2b. PMID 16601427